CLINICAL TRIAL: NCT07404059
Title: The Effect of Fat Cavitation Versus Pneumatic Compression on Adipose Tissue Thickness in Patients With Lipedema
Brief Title: Effect of Ultrasound Cavitation Versus Pneumatic Compression on Adipose Tissue Thickness on Lipedema Patients
Status: Available | Type: Expanded Access
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Sayed, Dr, Cairo University
Other Study IDs: lipedema
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lipedema
Keywords: pneumatic compression; fat cavitation; lipedema
MeSH Terms: conditions — Lipedema

INTERVENTIONS:
Device: fat cavitation — fat cavitation is a device produces ultrasound waves used for fat lipolysis

SUMMARY:
PURPOSE:

This study will be conducted to investigate any significant effect of ultrasound fat cavitation or pneumatic compression on adipose tissue thickness in patients with lipedema.

BACKGROUND:

Lipedema is a connective tissue disorder that cause physical discomfort and psychological stress.

A literature review published in 2020 estimated that 10-11% of women or approximately 400 million women across the globe have lipedema.

Lipedema fat is dangerous when it progress onto abdomen and trunk resulting in a risk of developing high blood pressure, high cholesterol and diabetes.

Ultrasound cavitation is a safe cosmetic procedure has almost no adverse reactions used to break down fat cells under the skin which improves the body shape and reduce circumference which make it a promising non invasive tool alternative to surgical liposuction.

Pneumatic compression is bl=elieved to reduce the limb circumference and volume which make it a good treatment option for lipedema.

HYPOTHESES:

Null Hypothesis:there will be no significant effect of fat cavitation or pneumatic compression on the adipose tissue thickness in patients with lipedema.

RESEARCH QUESTION:Will be any significant effect of fat cavitation or pneumatic compression on the adipose tissue thickness in patients with lipedema

DETAILED DESCRIPTION:
Lipedema is a progressive disease. There are currently 3 primary stages that describe disease severity: stage 1 involves thickening of subcutaneous tissue and disproportion accumulation of subcutaneous tissue in the extremities (tissue remains smooth and is generally not heavy or swollen); stage 2 is characterized by increased fibrous tissue, leading to a nodular feel in the subcutaneous tissue. Symptomatic lipedema patients at stage 2 and higher almost always have secondary swelling on physical exam and most with evidence of impaired lymphatic function. Stage 3 involves progression with the formation of lobules of skin and subcutaneous tissue Conservative therapies, including manual lymphatic drainage, compression therapy, decongestive sports/movement therapy, skin care, and empowerment are currently considered as first line treatments (2-4). Surgical reduction of pathological SAT with lymph-sparing liposuction in wet-technique is another potential therapeutic option to improve symptoms, mobility and overall quality of life The most promising techniques for noninvasive body sculpturing purposes are based on ultrasound-induced fat cavitation. Liporeductive ultrasound devices afford clinically relevant subcutaneous fat pad reduction without significant adverse reactions, noninvasive transcutaneous ultrasound cavitation is a promising and safe technology for localized reduction of fat and provides experimental evidence for its specific mechanism of action on the adipocytes. the most effective instruments for noninvasive fat reduction use ultrasounds through the generation of compression and depression cycles at appropriate frequency, they cause cavitation phenomena at the fat droplet-watery cytoplasm interface and eventually adipocyte rupture and triglyceride release. the thermal effects of focused ultrasound energy may result in adipocyte necrosis in the treatment area. The most recent devices for liporeductive purposes have been specifically designed to prevent unwanted tissue injury. a focused ultrasound emitter, was first demonstrated to achieve selective adipocyte lysis and clinically relevant reduction of the volume of subcutaneous fat pad, in the absence of significant adverse reactions.

Pneumatic compression devices move lymphatic fluid and support the elimination of proteinaceous fluids, thus leading to improved patient-reported symptoms, decreased limb girth and volume, increased elasticity of tissues, and fewer episodes of infection. Atan et al. found improvements in limb volume, pain, and physical functioning in patients with stage 3 or 4 lipedema after CDT or PCD treatmentSzolnoky reported daily treatment with CDT, PCD, and multilayered short-stretch bandaging performed for 5 days led to significant improvements in leg volume, capillary fragility, and pain in women with lipedema 90 patients will participate in the study for 3 months, and randomly be assigned into 3 equal groups. Study Group (A), (n =30) will receive fat cavitation 2 times /week for 3 months in addition to the complete decongestive therapy , study group (B), (n =30) will receive pneumatic compression 3-5 times /week in addition to the complete decongestive therapy, and control group (c), (n=30) will receive the complete decongestive therapy only.

Hypothesis:

This study will test the following hypothesis:

* There is no effect of cavitation on the adipose tissue thickness in patients with lipedema.
* There is no effect of pneumatic compression on adipose tissue thickness in patients with lipedema.

Basic assumption:

• It will be assumed that:

1. All patients will be free from any condition that may affect or delay the response to our program such as diabetes, open wound or hypertension.
2. The assessment methods will be valid and reliable.
3. All patient will be accurately diagnosed and exclude any other similar conditions as lymphedema, lipohypertrophy or Dercum's disease.
4. All patients will be cooperative during the assessment and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ninety females patients their age from 30 to 45 years
2. Diagnosed with mild to moderate lipedema
3. Mentally stable functionally and physically stable.

Exclusion Criteria:

1. Patents with severe lipedema
2. Patients with type 4 lipedema
3. Clinically unstable patients
4. Patients with chronic diseases
5. Patients with endocrine diseases
6. Patienst with similar conditions like lymphedema, dercum's diseases or overall obesity
7. Patients with lower limbs fractures

Ages: 30 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — females has lipedema as lipedema is affecting only females at periods of hormonal changes as puberty, pregnancy or menopause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt